CLINICAL TRIAL: NCT05267366
Title: Phase II Randomized Trial of Carboplatin/Cisplatin+Pemetrexed+PD-1 Inhibitor+/- Bevacizumab in Stage IV Non-squamous NSCLC
Brief Title: Chemotherapy Combines With Bevacizumab and PD-1 Inhibitor in Non-squamous NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qingdao Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QDCH2022-02-15
Record Dates: First submitted 2022-02-14; First posted 2022-03-04 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: PFS; OS
MeSH Terms: interventions — Immune Checkpoint Inhibitors; Bevacizumab; Carboplatin; Cisplatin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemothreapy with PD-1 inhibitor and bevacizumab (Experimental): PD-1 inhibitor (pembrolizumab) 200mg iv day 1 Carboplatin 5 AUC /cisplatin 75 mg/m2, iv day 1 Pemtrexed 500 mg/m2, iv day 1 Bevacizumab 15 mg/m2, iv day 1 as induction therapy every 21 days a cycle for 4 cycles, PD-1 inhibitor (pembrolizumab) 200mg iv day 1 Bevacizumab 15mg/m2, iv day 1 every 21 days a cycles as maintenance treatment for 31 cycles or 2 years.
  Interventions: Drug: PD-1 inhibitor, Bevacizumab, Carboplatin, Cisplatin, Pemtrexed
- Chemothreapy with PD-1 inhibitor (Active Comparator): PD-1 inhibitor (pembrolizumab) 200mg iv day 1 Carboplatin 5 AUC /cisplatin 75 mg/m2, iv day 1 Pemtrexed 500 mg/m2, iv day 1 as induction therapy every 21 days a cycle for 4 cycles, PD-1 inhibitor (pembrolizumab) 200mg iv day 1 every 21 days a cycles as maintenance treatment for 31 cycles or 2 years.
  Interventions: Drug: PD-1 inhibitor, Bevacizumab, Carboplatin, Cisplatin, Pemtrexed

INTERVENTIONS:
Drug: PD-1 inhibitor, Bevacizumab, Carboplatin, Cisplatin, Pemtrexed — PD-1 inhibitor (pembrolizumab) 200mg iv, d1; bevzcizumab 15mg/kg, iv, d1; Carboplatin 5/AUC or Cisplatin 75mg/m2 iv d1; Pemtrexed 500mg/m2 iv, d1; every 21 days a cycle.

SUMMARY:
In recent years, immunotherapy has emerged as a form of treatment that can lead to robust responses in a subset of patients. PD-1 inhibitor plus chemotherapy showed prolonged survival in NSCLC by the study of KEYNOTE 024, KEYNOTE 189 etc. Thus, this study combines immunotherapeutic agent PD-1 inhibitor with an ant-angiogenic agent, bevacizumab, and double platinum therapy (carboplatin/cisplatin and pemetrexed).

ELIGIBILITY:
Inclusion Criteria:

* • Must have histologically or cytologically confirmed stage IV non-squamous non-small cell lung cancer

  * Must have not harbor an EGFR mutation in exon 19 or exon 21, or without an ALK or ROS1 rearrangement,.
  * Must have measurable disease by CT or MRI, defined as at least one lesion that can be accurately measured in at least one dimension in accordance with RECIST criteria v 1.1
  * Age > 18 years
  * ECOG performance status of 0 or 1, or 2.
  * Must have normal organ and marrow function as defined below. The use of G-CSF should follow standard recommendations and physician discretion. If blood transfusion is performed for achieving hemoglobin levels, the levels should stay at ≥ 9.0 mg/ml for at least a week after transfusion.

Absolute neutrophil count > 1,500/mcL Hemoglobin ≥ 9.0 mg/ml Platelets > 100,000/mcL Total bilirubin ≤1.5 X institutional upper limit of normal (ULN) AST/ALT (SGOT/SGPT) < 3 times institutional normal limits, or up to 5 times institutional normal limits if the patient has liver metastases Creatinine OR Creatinine clearance ≤1.5 X ULN, OR > 40 Ml/min/1.73 m2 for patients with creatinine levels above institutional normal as per Cockcroft-Gault formula International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants Activated Partial Thromboplastin Time (aPTT) <1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants Thyroid stimulating hormone (TSH) Within normal limits a

a: If TSH is not within normal limits at baseline, the subject will still be eligible if total T3 or free T4 are within normal limits.

* Full-dose anticoagulation must be on a stable dose (minimum duration 14 days) of oral anticoagulant or low molecular weight heparin (LMWH). If receiving warfarin, the patient must have an INR ≤3.0. For heparin and LMWH there should be no clinically significant active bleeding (with no bleeding within 14 days prior to first dose of protocol therapy) or pathological condition present that carries a high risk of bleeding (for example, tumor involving major vessels or known varices).
* Ability to understand and willingness to sign a written informed consent and HIPAA consent document.
* A biopsy, either core, cell block from FNA or cell block from surgical resection, must be available for the study. If the sample is not adequate, the patient must agree to provide a fresh biopsy specimen before the start of treatment. Any available archival tissue will also be collected. While a biopsy sample must be adequate and available for the study, an inadequate tissue sample would not be explicitly exclusionary and further discussion with the sponsor is allowed to assess the eligibility of the patient for the trial if, for clinical or other reasons, a new biopsy sample cannot be obtained.
* Urinary protein must be ≤1+ on dipstick or routine urinalysis (UA; if urine dipstick or routine analysis is ≥2+, a 24 hour urine collection for protein must demonstrate <1000 mg of protein in 24 hours to allow participation in the protocol).

Exclusion Criteria:

* . Received prior therapies targeting PD-1, PD-L1, CTLA-4 or other immune checkpoints.

  * Received prior platinum-based chemotherapy for advanced disease.
  * Patients who have received prior systemic anti-vascular therapy (e.g., bevacizumab and small molecule VEGFR inhibitors) for advanced disease (Cohort 2)
  * Treatment with any approved systemic anti-cancer therapy or systemic immune-stimulatory agents (including but not limited to interferons, interleukin IL-, and tumor necrosis factor) within 28 days prior to initiation of study treatment.
  * Clinically uncontrolled pleural effusion or ascites that requires pleurocentesis or abdominal tapping for drainage within 2 weeks prior to initiation of study treatment.
  * Active leptomeningeal disease or uncontrolled brain metastasis.
  * History of allergic reactions to any study drugs.
  * CrCl < 45 mL/min
  * Patients with active viral hepatitis that requires treatment.
  * Active autoimmune diseases that requires treatment and may affect study treatment estimated by investigator.
  * Any condition that required systemic treatment with either corticosteroids or any other immunosuppressive medication that may affect study treatment estimated by investigator.
  * Severe chronic or active infections requiring systemic antibacterial, antifungal or antiviral therapy.
  * History of hemoptysis, i.e., coughing up at least one-half teaspoon of fresh blood, within 3 months prior to enrollment. (Cohort 2)
  * Imaging shows tumor invasion of a large vessel (e.g., pulmonary artery or superior vena cava) that the investigator determines is at risk for bleeding. (Cohort 2)
  * Had minor surgical procedures, such as tube placement, within 48 hours prior to first bevacizumab treatment. (Cohort 2)
  * Recently treated with a full dose oral or parenteral anticoagulant or thrombolytic agent. Prophylactic using anticoagulants is allowed. (Cohort 2)
  * History or test results indicating an inherited bleeding tendency or coagulation disorder that may increase the risk of bleeding (cohort 2)
  * uncontrolled hypertension (systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg) (cohort 2)
  * Clinically meaningful (e.g., active) cardiovascular disease that, in the judgment of the investigator, is intolerant to bevacizumab therapy (cohort 2)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | up to 24 months
  Progression-free survival (per RECIST 1.1) is defined as the time from the starting date of study drug to the date of first documentation of disease progression or death, whichever occurs first.
Overall Survival (OS) | up to 24 months
  OS is defined as the time from the starting date of study drug to the date of death due to any cause.

SECONDARY OUTCOMES:
Objective Respond Rate (ORR) | up to 24 months
  ORR (per RECIST 1.1) is defined as the proportion (%) of patients with at least one visit response of complete response (CR) or partial response (PR).
Duration of Response (DoR) | up to 24 months
  DoR (per RECIST 1.1) is defined as the time from the date for first documented response of complete response (CR) or partial response (PR) to the date of first documented of disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Qingdao central Hospital, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No